CLINICAL TRIAL: NCT05491486
Title: The Relationship Between Mindfulness and Empathy With the Oxytocinergic System in Persons With Schizophrenia
Brief Title: Mindfulness, Empathy and the Oxytocinergic System in Persons With Schizophrenia
Acronym: OXYGEN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Principal Investigator, Kerem Böge, Dr. Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OXYGEN2022
Record Dates: First submitted 2022-08-03; First posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Schizophrenia Spectrum and Other Psychotic Disorders
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: The condition will be revealed to the participants after all T0 assessments have been completed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based Group Therapy (MBGT+TAU) (Experimental): Participants randomized into the experimental condition attend MBGT for four weeks in addition to regular university hospital outpatient treatment as usual (TAU). Overall, the core modules of the program are based on mindfulness-based cognitive therapy, taking into account both Chadwick's recommendations for implementing mindfulness in psychosis as well as patient feedback. Each week, a new topic is introduced to enhance the understanding of four core aspects of mindfulness (breath, senses, detachment, and body awareness). The therapy sessions will be held by a psychotherapist in training in cognitive behavioral therapy with over three years of experience in mindfulness practice and supervised by a psychotherapist with more than a decade of experience in mindfulness-based therapeutic approaches. Within the sessions, short periods of meditation are used to avoid prolonged periods of silence, and basic anchoring techniques and easy-to-understand language are used.
  Interventions: Behavioral: Mindfulness-based Group Therapy
- Treatment as Usual (No Intervention): All participants will be recruited from the outpatient facility at the Charité - Universitätsmedizin Berlin, Campus Benjamin Franklin and therefore, the heterogeneity of the obtained treatment options can be limited. As the standard procedure in our outpatient facility, patients will be seen monthly by a psychiatrist as well as individual sessions by a psychotherapist or psychiatric nurse (1:2 ratio). Hence, regardless of the study condition, all participants will obtain high standard health care at a renowned university hospital outpatient facility according to official national and international treatment guidelines providing pharmacological therapy, psychological consultation, and, on-demand, psychosocial support by social workers. The amount of psychotherapy received and on-demand psychosocial support will be recorded during the study period.

INTERVENTIONS:
Behavioral: Mindfulness-based Group Therapy — see above
  Arms: Mindfulness-based Group Therapy (MBGT+TAU)

SUMMARY:
Recent studies indicated positive effects of mindfulness-based interventions (MBI) for schizophrenia (SCZ), but also on oxytocin (OXT) levels in healthy persons. It was also shown that response to MBI could be shaped by genetic factors. However, the interplay between mindfulness and empathy and genetic factors with the oxytocinergic system has not yet been examined in SCZ. The aim of the current explorative study is to (1) explore the effect of mindfulness-based group therapy (MBGT) on OXT levels as well as empathy in persons with SCZ; (2) investigate whether polygenic risk scores (PRS) for empathy can predict empathy levels in persons with SCZ; (3) investigate whether PRS for empathy and specific genetic configurations in the oxytocin receptors are associated with MBGT outcomes and OXT levels; 4) examine changes in positive- and negative symptoms, depression, anxiety, social functioning, and mindfulness at a within-group level and between both conditions.

A parallel-group, proof-of-concept randomized controlled trial with 30 participants allocated to each trial arm (N = 60) will be conducted. Participants will be randomly assigned to MBGT alongside treatment as usual (MBGT+TAU) or treatment as usual (TAU). For a treatment period of four weeks, participants will receive weekly MBGT sessions. Four weeks after baseline assessments (T0), post-intervention assessments (T1) will take place. As a pilot study, effect sizes will be estimated for within- and between-group effects with corresponding confidence intervals.

Outcomes of our proof-of-concept study can provide insight into potential biological mechanisms underlying mindfulness in SCZ, determine a valid biomarker associated with empathy and negative symptoms and pave the way for a personalized treatment approach for individuals with SCZ.

ELIGIBILITY:
Inclusion Criteria:

* be aged between 18 and 65
* meet diagnostic criteria for schizophrenia (ICD-10: F20.X) ascertained by a trained psychiatrist
* sufficient German language proficiency to engage with the intervention
* no recent (<4 weeks) major change in psychopharmacologic medication
* be able to give written informed consent

Exclusion Criteria:

* a score of 7 on any item of the positive scale of PANSS, suggesting severe psychotic symptoms
* acute suicidality
* current substance use other than nicotine
* neurological disorders or brain damages

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-07-15 (Estimated); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
Change in oxytocin levels | Baseline and week 4
  Venous blood samples will be taken to determine the basal oxytocin plasma to obtain an individual baseline and comparison level. Furthermore, saliva samples will be taken before and after each MBGT session to determine OXT levels.
Change in empathy levels IRI | Baseline and week 4
  Interpersonal Reactivity Index (IRI)
  The IRI measures empathy on four subscales: perspective taking, fantasy, empathic concern and personal distress. Each subscale consists of 4 items rated on a 7-point Likert scale. The internal consistent is satisfactory with a Cronbach´s alpha of .78.
Change in empathy levels EQ | Baseline and week 4
  Empathy Quotient (EQ)
  The EQ consists of 40 statements to which participants have to indicate the degree to which they agree or disagree. There are four response options: 'strongly agree', 'slightly agree', 'slightly disagree', 'strongly disagree'. 'Definitely agree' responses score two points and 'slightly agree' responses score one point on half the items, and 'definitely disagree' responses score two points and 'slightly disagree' responses score one point on the other half. The remainder of the response options score 0.
  Finally, Cronbach's alpha was 0.92, which is high.

SECONDARY OUTCOMES:
Change in SMQ Mindfulness | Baseline and week 4
  The SMQ comprises 16 items that are rated on a seven-point Likert-scale ranging from (6) "agree totally" to (0) "disagree totally". Consequently, the total score ranges from 0 to 96, with a higher score indicating higher mindfulness. The internal consistency of the German version of the SMQ was Cronbach's α = 0.89.
PSP Social Functioning | Baseline
  The Personal and Social Performance Scale (PSP) is a rater-based questionnaire used to assess social functioning in patients with SSD. The PSP showed good test-retest reliability (ICC = 0.79) in patients with schizophrenia
Change in PANSS Positive, Negative, and General Symptoms | Baseline and week 4
  The Positive and Negative Syndrome Scale (PANSS) is one of the most widely used rater instruments for the assessment of the presence and severity of psychotic symptoms. Each scale comprises seven statements which are rated by the interviewer using a seven-point Likert format (from 1= absent to 7= extreme). The PANSS is reported to have satisfactory internal consistency, good interrater reliability and construct validity.
Change in SNS Negative Symptoms | Baseline and week 4
  This is a 20-item self-reported questionnaire with five subscales, namely alogia, avolition, anhedonia, social withdrawal and diminished emotional range. These subscales cluster on two factors, the apathy and emotional components. Participants can estimate the answer to each question on a scale from 0 (strongly disagree) to 3 (strongly agree). The scale was shown to have good internal consistency with Cronbach's alpha = .87.
Change in DASS Depression & Anxiety | Baseline and week 4
  The 21-item Depression, Anxiety, and Stress Scale (DASS-21) is assessed on a four-point Likert-scale ranging from (0) "did not apply to me at all over the last week" to (3) "applied to me very much last week." It shows internal consistencies of α > 0.80 across the three subscales and has shown to be a useful measurement tool for patients with SSD.
Change in CFQ Psychological Flexibility | Baseline and week 4
  The instrument is self-reports, which showed high internal consistency in previous studies.
Change in PANAS Positive and Negative Affect | Baseline and week 4
  The PANAS contains 20 items, each consisting of an adjective describing an emotion. The participants have to select how applicable this adjective is to their current state from 1 (not at all) to 5 (extremely). Ten items are assigned to the positive (e.g. "Excited") as well as the negative scale (e.g. "Fearful"). The reliability of the PANAS ranges from .86 to .93.
Change in BIRT Motivation (BMQ) | Baseline and week 4
  The BIRT Motivation Questionnaire comprises 34 statements rated on a 4-point likert scale (always, often, sometimes, never). Internal consistencies of the BMQ-S and BMQ-R were high (Cronbach's alpha=.94 & .95 respectively).

OTHER OUTCOMES:
Polygenic Risk Scores (PRS) | Baseline
  We investigate whether polygenic risk scores (PRS) for empathy can predict empathy scores across groups at baseline in individuals with schizophrenia. For this purpose, the subject's genotypes will be examined. PRS have been shown to be associated with complex genetic traits such as empathy and mental disorders such as schizophrenia or autism spectrum disorders. Moreover, we will investigate whether empathy-PRSs and specific genetic configurations in the OXTR are associated with MBGT outcomes and OXT levels in blood samples on an exploratory level.

CONTACTS AND LOCATIONS:
Locations (1):
- Charité - Universitätsmedizin Berlin, Campus Benjamin Franklin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No